CLINICAL TRIAL: NCT04653441
Title: Resilience-based Psychosocial Intervention Among Children Affected by HIV/AIDS in China
Brief Title: Resilience-based Psychosocial Intervention Among Children Affected by HIV/AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Henan University (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Xiaoming Li, Professor and Endowed Chair, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00047860
Record Dates: First submitted 2019-03-06; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Emotional Adjustment; Aids/Hiv Problem
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: The proposed multimodal "Child Caregiver-Advocacy-Resilience" intervention (ChildCARE) will include three integrated components: the individual child (peer-group activities), family (caregiver parenting skill training), and the local community (community advocacy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Child-only Intervention (Experimental): The children in this arm will receive only child intervention curriculum (peer group activities). The child intervention includes 20 hours of facilitator-guided programming delivered in 10 sessions in a peer-group setting and aims to increase resilience by developing a number of skills including positive thinking, emotional regulation, coping, and problem solving.
  Interventions: Behavioral: Child-Caregiver-Advocacy-Resilience [ChildCARE] intervention
- Child+Caregiver Intervention (Experimental): The children in this arm will receive child intervention and their caregivers will receive the caregiver intervention, At the caregiver level, caregivers receive 10 hours of facilitator-guided programming delivered in five sessions that aims to increase positive parenting skills and build the capacity of the caregiver to engage in self-care and seek support.
  Interventions: Behavioral: Child-Caregiver-Advocacy-Resilience [ChildCARE] intervention
- Child+Caregiver+Community Intervention (Experimental): The children in this arm will received child intervention; their family will receive caregiver intervention and community-based intervention. At the community level, trained community advocates (e.g., teachers, village nurses) conduct monthly home visits and organize a series of community-based activities over a period of two years to promote cohesion and strength within local communities and to increase community support for affected families.
  Interventions: Behavioral: Child-Caregiver-Advocacy-Resilience [ChildCARE] intervention
- Attention Control (No Intervention): Children and caregivers who do not receive any intervention activities

INTERVENTIONS:
Behavioral: Child-Caregiver-Advocacy-Resilience [ChildCARE] intervention — The proposed multimodal "Child Caregiver-Advocacy-Resilience" intervention (ChildCARE) will include three integrated components: the individual child (peer-group activities), family (caregiver parenting skill training), and the local community (community advocacy).
  Arms: Child+Caregiver Intervention; Child+Caregiver+Community Intervention; Child-only Intervention

SUMMARY:
Parental illness and death from HIV/AIDS has a profound and lasting impact on a child's psychosocial well-being, potentially challenging the basic needs for survival and compromising the child's future. Therefore, the impact of parental HIV/AIDS on children needs to be treated from both a public health and a developmental perspective. However, to date the role of a resilience-based approach among children affected by HIV is hypothesized but not evidence-based. In this application, we propose to develop a theory-guided, resilience-based, multimodal intervention by culturally adapting and integrating components from three SAMHSA model programs which show strong evidence in promoting protective factors among young children. The multimodal intervention will include three approach levels: the individual child (peer-group activities), the family (caregiver parenting skill training), and the local community (community advocacy). The short, medium, and long-term efficacy of the Child-Caregiver-Advocacy-Resilience [ChildCARE] intervention to improve health and psychosocial well-being of children will be evaluated over 36 months through a cluster randomized controlled trial. About 800 HIV/AIDS-affected children (8 to 11 years of age) and their primary caregivers will be recruited from central China where we have built a strong research infrastructure and community collaboration during our previous study. The primary outcome measures for the children will include physical health, mental health, growth and development, school performance, and a biological indicator of neurobiological stress response (salivary cortisol). The outcome measures at caregiver level will include parenting style, parental engagement, and mental health well-being. The changes at the community level will be measured using children's and caregivers' perceptions of social support and HIV-related public stigma. We will also examine the potential mechanism through which the ChildCARE intervention is exerting its impact by identifying improvement in protective factors and other individual and contextual factors that potentially mediate or moderate the intervention effect. This proposed project will examine whether the multilevel protective factors we identified in our initial project are amenable to intervention and whether their hypothesized changes explain improvement in children outcomes.

DETAILED DESCRIPTION:
During the past five years (09/05-08/10) we were funded by R01MH76488 to study the psychosocial needs of children affected by HIV including both orphans (children under 18 who lost one or both of their parents to HIV/AIDS) and vulnerable children (children with one or both parents infected with HIV) in rural China. The overarching goal of our previous study was to inform the development of effective, culturally appropriate, and sustainable psychosocial interventions for these children. Guided by a developmental psychopathology perspective, we constructed an assessment model that integrated research findings from the literatures on bereavement, attachment, risk and resilience to delineate the children's psychosocial needs following HIV-related parental death or illness1. We incorporated both individual and environmental factors that potentially could moderate or mediate the negative effects of parental HIV/AIDS on these children. The comprehensive qualitative and quantitative data we collected and reported in 29 peer-reviewed publications during the past five years have provided the critical foundation for a cultural adaptation of theory-driven psychosocial prevention programs among children affected by HIV. The main findings from this body of research included 1) children affected by HIV experienced greater mental and developmental challenges (e.g., trauma symptoms, depression, social isolation, poor school performance) than comparison children who were from the same community but did not experience HIV-related illness and death in their families; 2) some children demonstrated tremendous resilience reflected in good school performances and the absence of elevated levels of psychosocial problems despite parental HIV/AIDS and other traumatic events in their lives; and, 3) key protective factors exist within the child and the social environment (e.g., positive future orientation, trusted caregivers, and supportive community) which could contribute to resilience in these children, and hence buffer the children from the detrimental effects of parental HIV/AIDS. The proposed project will examine whether the protective factors identified in our previous study are amenable to intervention and whether their hypothesized changes can indeed explain improvement in mental and developmental outcomes among participating children.

From research on early childhood development, compelling evidence has revealed the critical importance of successful adaptation in the face of adversity ("resilience") for laying the foundation for successful adjustment later in life2-4. However, to date the utility of a resilience-based intervention approach among children affected by HIV is hypothesized but not evidence-based5-6.Therefore, in this application, we propose to adapt three evidence-based programs to produce a theory-driven resilience-based intervention to improve the well-being of children affected by HIV in rural China. The proposed multimodal "Child Caregiver-Advocacy-Resilience" intervention (ChildCARE) will include three integrated components: the individual child (peer-group activities), family (caregiver parenting skill training), and the local community (community advocacy). The short, medium, and long-term efficacy of the ChildCARe intervention will be evaluated over 36 months through a cluster randomized controlled trial (RCT). The primary outcome measures for the children will include physical health, mental health, growth and development, school performance, and a biological indicator of neurobiological stress response (i.e., salivary cortisol). There are three specific aims and four hypotheses in our application:

AIM #1: Develop a theory-guided, resilience-based, multimodal intervention [ChildCARe] by culturally adapting and integrating components from three SAMHSA model programs which show strong evidence in promoting protective factors among children; the adaptation process will be informed by 1) the data collected from our previous study; 2) our 18 years' experience in developing and adapting effective HIV behavioral prevention programs in various cultural settings including China; and 3) input from the local collaborators and communities (e.g., community advisory board and research participants); AIM #2: Test the efficacy of the ChildCARe intervention through a cluster RCT involving 800 HIV-affected children (8 to 11 years of age) and their primary caregivers from 80 villages in central China where we have built a strong research infrastructure and community collaboration during our previous study; AIM #3: Examine the potential mechanism of the intervention by identifying improvement in protective factors and other individual and contextual factors that potentially mediate or moderate the intervention effect;

Hypothesis #1: The ChildCARe intervention will demonstrate short, medium, and long-term efficacy in improving children's primary outcomes and biological indicator (salivary cortisol); Hypothesis #2: The ChildCARE intervention will demonstrate short, medium, and long-term efficacy in improving children's intermediate outcomes (e.g., social-emotional competence, positive future orientation, and trusting relationship with current caregivers), caregiver's outcomes (e.g., parenting skills, mental health well-being), and community-level outcomes (e.g., children's and caregivers' perceptions of social support); Hypothesis #3: Improvement in intermediate outcomes at levels of child, family, and community will mediate the effect of the ChildCARE intervention on the children's primary outcomes and biological indicator; Hypothesis #4: Some contextual factors (e.g., care arrangement, household socioeconomic status [SES], caregiver's physical health status, disease progression for caregivers living with HIV) will moderate the effect of ChildCARE intervention on the children's primary outcomes and biological indicator.

ELIGIBILITY:
Inclusion Criteria:

* 8 to 17 years of age
* having lost one or both parent to AIDS (orphans) or are currently living with a HIV-positive parent (vulnerable children)

Exclusion Criteria:

* children living in centralized care setting;
* known HIV-infection;
* physical illness and developmental disability (e.g., severe mental retardation) that prevent them from engaging routine daily activities;
* plan to permanently relocate outside of the province within a year.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 790 (Actual)
Dates: Start 2011-09-15 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
change of psychological resilience at 36 months follow up | 7 waves during 36 months with a 6-month interval
  Resilience-related outcomes at child level
change of school performance at 36 months follow up | 7 waves during 36 months with a 6-month interval
  Children's academic performance and other schooling outcomes
change of mental health status at 36 months follow up | 7 waves during 36 months with a 6-month interval
  Children's mental health outcomes

SECONDARY OUTCOMES:
change of parenting practices at 36 months follow up | 4 waves (from caregivers) over 36 months
  perceptions and practices of parenting reported by both children and caregivers
Changes of parental depression at 36 months follow up | 4 waves over 36 months
  Caregiver mental health outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Li, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li X, Harrison SE, Fairchild AJ, Chi P, Zhao J, Zhao G. A randomized controlled trial of a resilience-based intervention on psychosocial well-being of children affected by HIV/AIDS: Effects at 6- and 12-month follow-up. Soc Sci Med. 2017 Oct;190:256-264. doi: 10.1016/j.socscimed.2017.02.007. Epub 2017 Feb 13. PMID 28215430